CLINICAL TRIAL: NCT02029092
Title: BIOTRONIK- Safety and Performance Registry for an All Comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice III- ELADIS
Brief Title: BIOFLOW III Satellite-ELADIS Orsiro Stent System
Status: Completed | Type: Observational
Sponsor: C.E.M. Biotronik, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: G1302
Record Dates: First submitted 2013-12-19; First posted 2014-01-07 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: International; Multicenter; Observational registry; Orsiro Drug Eluting Stent (DES); Stenting; Treatment of coronary artery disease; Coronary revascularization; Percutaneous Coronary Intervention (PCI); STEMI; NSTEMI; Ischemia; Angina; Acute Myocardial Infarction (AMI); Small Vessels; Chronical Total Occlusion (CTO)
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro

SUMMARY:
This registry is a clinical evaluation of the Orsiro LESS in subjects requiring coronary revascularization with Drug Eluting Stents (DES). It is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD) treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedure success. However, the medium to long-term complications range from rather immediate elastic coil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30 to 50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in De Novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20 to 40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neontimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

Therefore this observational registry has been designed for the clinical evaluation of the ORSIRO LESS requiring coronary revascularization with DES. Results will contribute to the collection of clinical evidence for the clinical performance and safety of ORSIRO drug eluting stent system in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is≥18 years of age.

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation, antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media.
* Planned surgery within 6 months after PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not yet reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects requiring coronary revascularization with Drug Eluting Stents (DES)
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
TLF | 6 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR).
Target Vessel Revascularization (TVR) | 6 and 12 months
  Target Vessel Revascularization (TVR)
Target lesion revascularization (TLR) | 6 and 12 months
  Target lesion revascularization (TLR)
Stent Thrombosis rate | 6 and 12 months
  Stent Thrombosis rate
Device success | up to discharge
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation, without using any adjunctive device outside the assigned treatment strategy
Procedure success | up to 7 days after procedure
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation, without using any adjunctive device and without the occurrence of ischemia-driven major cardiac event during the hospital stay to a maximum of the first seven days post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Martin, Study Director — CEM BIOTRONIK SA
Locations (14):
- Spain (14):
  - Hospital Universitario León, León, A/Altos de Nava S/n
  - Hospital Infanta Cristina, Badajoz
  - Hospital Vall D' Hebron, Barcelona
  - Hospital G.de Jerez de la Frontera, Cadiz
  - Hospital de Mérida, Mérida
  - Hospital Univ. Virgen de la Arrixaca, Murcia
  - Hospital Parc Tauli, Sabadell
  - Complejo de Hospitalario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Clinico de Valencia, Valencia
  - Hospital Doctor Peset, Valencia
  - Hospital de Txagorritxu, Vitoria-Gasteiz
  - Hospital de Cruces, Vizcaya